CLINICAL TRIAL: NCT04627688
Title: Optimization of Diet Before Surgery (OptiSurg): Effects of Time Restricted Feeding (TRF) Before Vascular Surgery - An Open-label Randomized Controlled Trial of TRF vs Regular Dietary Advices
Brief Title: Optimization of Diet Before Surgery (OptiSurg)
Acronym: OptiSurg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Alban Longchamp, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-02483
Record Dates: First submitted 2020-10-19; First posted 2020-11-13 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Surgery; Time Restricted Feeding
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dietary advices (Active Comparator)
  Interventions: Behavioral: Standard dietary advices
- Time restricted feeding (Experimental)
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will be advised to eat only during a selected window of 8 hours, and no later than 4pm, with no advice on nutrition quality, quantity or caloric intake. The intervention will include no medication, no medical device, and will last for 2 weeks prior to surgery.
  Arms: Time restricted feeding
Behavioral: Standard dietary advices — Participants will be given standard dietary advices, as recommended by the international nutrition guidelines, and thus are not different from common clinical practice.
  Arms: Standard dietary advices

SUMMARY:
The overarching goal of this project is to assess whether a controlled short-term Time restricted feeding (TRF) intervention leads to metabolic benefits, improves recovery after vascular surgery and that TRF is safe. Participants suffering from intermittent claudication (Fontaine stage II peripheral artery disease, PAD) will be randomly assigned to a 2-week TRF or active control dietary advices before open surgical revascularization. Prior to the surgery, the investigators will assess the eating patterns of participants with an innovative smartphone application ('app') which is less intrusive and more reliable than food diaries/questionnaires to assess eating behavior and patterns. In the second part of the study, the investigators will investigate whether a short term TRF intervention improves surgical recovery, in the short-term (1 month, primary endpoint) and long-term (optional, up to 1 year), as part of the routine clinical follow-up. This proposal builds on established expertise in the biology of dietary intervention, surgery, and study of eating patterns in human.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Fontaine stage II peripheral artery disease planned for open femoral endarterectomy
* Body mass index ≥ 20 kg/m2
* Smartphone compatible with the app (iOS or Android systems)
* Hypertensive (or on 1 or more blood pressure lowering medication)
* Hypercholesterolemia (or on 1 or more lipid lowering medication)

Exclusion Criteria:

* Diabetes on insulin therapy or sulfonylureas
* Fontaine stage III and IV peripheral artery disease
* Prior revascularization on the index leg within 14 days of the qualifying revascularization.
* Major surgery in the past 3 months
* Myocardial infarction or revascularization (PTA, stent, CABG) in the past 3 months
* Major illness / fever over the previous month, active cancer
* On a diet / weight management or prior bariatric surgery
* Major mental illness, unable to give consent, inability to follow study procedures (language barrier, dementia)
* Current shift work or travel abroad planned in the next month
* Major sleep disorder
* Enrolled in another interventional clinical trial
* Ongoing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with: Death, Myocardial infarction, Stroke, Surgical re-intervention. | 1 month
  Safety of TRF before vascular surgery

SECONDARY OUTCOMES:
Length of Stay [days] | 1 month
Change in systolic and diastolic blood pressure [mmHg] | 1 month
Change in ankle and toe brachial index [0.2-1.4] | 1 month
  Improvement in limb perfusion measured as an increase in the reported index
Change in weight [gram] | 1 month
Change in BMI [kg/m^2] | 1 month
Change in total cholesterol levels [mg/dl] | 1 month
Change in LDL cholesterol levels [mg/dl] | 1 month
Change in HDL cholesterol levels [mg/dl] | 1 month
Change in triglyceride levels [mg/dl] | 1 month
Change in glycemia [mmol/L] | 1 month
Change in insulin levels [pmol/L] | 1 month
Change in HbA1c levels [%] | 1 month
Adherence to TRF intervention | 1 month
  Adherence will be determined using the smartphone app, by the number of days in which a participant will be adherent to logging and all caloric food items were contained within a 15-min buffer on each side of the selected eating window.
Time from randomization to the first occurrence of any of the following major thrombotic vascular events: MI (Myocardial infarction), ischemic stroke, CV (Cardiovascular) death, ALI (Acute limb ischemia), and major amputation or death (any cause). | 1 year

OTHER OUTCOMES:
Change in interleukin-6,-1, -10 levels [pg/ml] | 1, 2 days ans 1 month
Change in tumor necrosis factor alpha levels [pg/mL] | 1, 2 days ans 1 month
Change in transforming growth factor beta levels [ng/mL] | 1, 2 days ans 1 month
Change in interferon gamma levels [pg/mL] | 1, 2 days ans 1 month
Change in cortisol levels [nmol/L] | 1, 2 days ans 1 month
Change in thyroid stimulating hormone levels [mIU/L] | 1, 2 days ans 1 month
Change in triiodothyronine levels [nmol/L] | 1, 2 days ans 1 month
Change in thyroxine levels [μg/d] | 1, 2 days ans 1 month
Change in circulating hydrogen sulphide levels | 1, 2 days ans 1 month
Change in circadian hormone secretion | 1, 2 days ans 1 month
Change in gut microbiome | 1, 2 days ans 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided